CLINICAL TRIAL: NCT06580548
Title: A New At-home Telerehabilitation Care Service Delivery Model for Stroke Survivors in the Rio Grande Valley
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Fadi Musfee, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-SPH-24-0166; 1UM1TR004906 (NIH)
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Stroke
Keywords: long-term rehabilitation management; stroke survivor; telehealth
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- CHW-supported telerehabilitation plus Usual Care (Experimental)
  Interventions: Device: CHW-supported telerehabilitation; Other: Usual Care

INTERVENTIONS:
Device: CHW-supported telerehabilitation — Participants will receive the Mobile Rehab mobile software, which allows participants to be prescribed personalized rehabilitation strengthening video regimens electronically based on respondent-indicated mobility and activities of daily living functionality
Other: Usual Care — Participants will be provide a list of local social services resources, including mental health, that participants can use . A callback number will be provided if they have any questions about the services.

SUMMARY:
The purpose of this study is to investigate the feasibility of a mobile telerehabilitation software for post-acute stroke care for Rio Grande Valley (RGV) stroke survivors with community health worker (CHW) at-home support and to estimate the functional health, mental health (depression), and caregiver burden outcomes of this new CHW-supported, at-home rehabilitation service delivery model and to identify salient barriers to and facilitators of adopting and delivering the new rehabilitation delivery model to further disseminate the model in real-world communities.

ELIGIBILITY:
Inclusion Criteria:

* A resident of the Brownsville, Texas (Cameron County) area
* SINGLE and FIRST qualifying stroke event with the ability to enroll and begin study activities within 3 months of onset of stroke event
* Pre-stroke modified Rankin score of ≤3 (less than moderate disability at baseline)
* Currently uninsured
* Spanish or English speaker
* Able to follow instructions (without aphasia that interferes with following instructions)
* Safe to perform basic strengthening rehabilitation exercises
* Able to stand with or without assistance

Exclusion Criteria:

* Aphasia or cognitive impairment (e.g., dementia) that interferes with following instructions or prevents following the study-related activities)
* Pre-stroke motor deficits
* Current psychiatric disorders, including substance use disorder
* Underlying brain pathologies inclusive of brain malignancies, multiple sclerosis
* Insured patients as insured patients are referred for standard-of-care clinical rehabilitation.
* Medical instability to participate in basic strengthening rehabilitation exercises
* Inability to access internet from home to access at-home rehabilitation software for intervention arm participants
* Having received any outpatient rehabilitation services prior to study enrollment for intervention arm participants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in basic mobility as assessed by the Acute Measure for Post-Acute Care (AM-PAC) Basic Mobility Outpatient Form (routine) | Baseline (week 1), week 3 (intervention participants only), week 6
  This is an 18 item questionnaire and each is scored from 1(unable) to 4( none) for a score range of 1-72, higher score indicating better outcome
Change in basic mobility as assessed by the Acute Measure for Post-Acute Care (AM-PAC) Basic Mobility Outpatient Form (low function ) | Baseline (week 1), week 3 (intervention participants only), week 6
  This is a 19 item questionnaire and each is scored from 0(unable) to 3( none) for a score range of 0-57, higher score indicating better outcome
Change in basic activity as Acute Measure for Post-Acute Care (AM-PAC) Daily Activity Outpatient Short Form (routine) | Baseline (week 1), week 3 (intervention participants only), week 6
  This is a 15 item questionnaire and each is scored from 1(unable) to 4( none) for a score range of 1-60, higher score indicating better outcome
Change in basic activity as Acute Measure for Post-Acute Care (AM-PAC) Daily Activity Outpatient Short Form (low function) | Baseline (week 1), week 3 (intervention participants only), week 6
  This is a 12 item questionnaire and each is scored from 0(total) to 3( none) for a score range of 1-36, higher score indicating better outcome
Change in Health-related quality of life as assessed by the European Health-Related Quality of Life- 5 Dimensions (EQ-5D) EuroQoL-5D five-level survey (EQ-5D-5L) | Baseline, week 3 (intervention participants only), week 6
  This is scored across 5 dimensions , mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and each dimension is scored on a five-level severity ranking that ranges from 1 (no problems) to 5 (extreme problems), higher score indicating worse outcome
Change in Depression as assessed by the Patient Health Questionnaire 9 (PHQ-9) | Baseline, week 3 (intervention participants only), week 6
  This is a 9 item questionnaire and each is scored from 0(not at all) to 3(nearly every day) for a score range of 0-27, higher score indicating worse outcome
Change in caregiver burden as assessed by the Zarit Burden Interview | Baseline, week 3 (intervention participants only), week 6
  This is a 12 item questionnaire and each is scored from 0(never) to 4(nearly always) for a score range of 0-48, higher score indicating worse outcome

SECONDARY OUTCOMES:
Acceptability/Appropriateness of the intervention for the stroke survivors as assessed by the Quantitative Implementation Measures for Stroke Survivors questionnaire | Baseline
  This is an 8 item questionnaire and each is scored from 1( strongly disagree) to 5(strongly agree) for a score range of 1-40, higher score indicating better outcome
Acceptability/Appropriateness of the intervention for the stroke survivors as assessed by the Quantitative Implementation Measures for Stroke Survivors questionnaire | week 7
  This is an 8 item questionnaire and each is scored from 1( strongly disagree) to 5(strongly agree) for a score range of 1-40, higher score indicating better outcome
Adoption of the intervention for the stroke survivors as assessed by the Quantitative Implementation Measures for Stroke Survivors questionnaire | Baseline
  This is an 5 item questionnaire and each is scored from 1( strongly disagree) to 5(strongly agree) for a score range of 1-25, higher score indicating better outcome
Adoption of the intervention for the stroke survivors as assessed by the Quantitative Implementation Measures for Stroke Survivors questionnaire | week 7
  This is an 5 item questionnaire and each is scored from 1( strongly disagree) to 5(strongly agree) for a score range of 1-25, higher score indicating better outcome
Acceptability & Appropriateness of the intervention for the community health workers as assessed by the Quantitative Implementation Measures for Community Health Worker questionnaire | Baseline
  This is an 7 item questionnaire and each is scored from 1( strongly disagree) to 5(strongly agree) for a score range of 1-35, higher score indicating better outcome
Acceptability & Appropriateness of the intervention for the community health workers as assessed by the Quantitative Implementation Measures for Community Health Worker questionnaire | week 7
  This is an 7 item questionnaire and each is scored from 1( strongly disagree) to 5(strongly agree) for a score range of 1-35, higher score indicating better outcome
Adoption of the intervention for the community health workers as assessed by the Quantitative Implementation Measures for Community Health Worker questionnaire | Baseline
  This is an 4 item questionnaire and each is scored from 1( strongly disagree) to 5(strongly agree) for a score range of 1-20, higher score indicating better outcome
Adoption of the intervention for the community health workers as assessed by the Quantitative Implementation Measures for Community Health Worker questionnaire | week 7
  This is an 4 item questionnaire and each is scored from 1( strongly disagree) to 5(strongly agree) for a score range of 1-20, higher score indicating better outcome
Feasibility of Community Health Worker as assessed by the Quantitative Implementation Measures for Community Health Worker questionnaire | Baseline
  This is an 7 item questionnaire and each is scored from 1( strongly disagree) to 5(strongly agree) for a score range of 1-35, higher score indicating better outcome
Feasibility of Community Health Worker as assessed by the Quantitative Implementation Measures for Community Health Worker questionnaire | week 7 (immediately after intervention)
  This is an 7 item questionnaire and each is scored from 1( strongly disagree) to 5(strongly agree) for a score range of 1-35, higher score indicating better outcome
Feasibility as assessed by the number of participants enrolled | end of study (week 7)
Adherence as assessed by the number of rehab videos watched in a day | end of study (week 7)
  adherence is defined by ≥1 daily mobile rehab video usage
Number of participants that view ≥1 daily mobile rehab videos | end of study (week 7)

CONTACTS AND LOCATIONS:
Overall Officials: Fadi Musfee, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States